CLINICAL TRIAL: NCT02163122
Title: A Pilot Study to Compare Responses to Cat Allergen Exposure Using the Environmental Exposure Chamber (EEC) and Nasal Allergen Challenge (NAC)
Brief Title: Cat Pilot Study - Environmental Exposure Chamber (EEC) vs. Nasal Allergen Challenge (NAC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DAIT ITN061AD
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Hypersensitivity, Immediate
Keywords: Cat Allergy; Feld1
MeSH Terms: conditions — Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NAC Followed by EEC (Experimental): This arm will undergo allergy assessment first by NAC. After a rest and washout period, the same individuals will undergo assessment in an EEC.
  Interventions: Procedure: Nasal Allergen Challenge; Other: Environmental Exposure Chamber; Biological: Cat allergen (FelD1)
- EEC Followed by NAC (Experimental): This arm will undergo allergy assessment first in an EEC. After a rest and washout period, the same individuals will undergo assessment by NAC.
  Interventions: Procedure: Nasal Allergen Challenge; Other: Environmental Exposure Chamber; Biological: Cat allergen (FelD1)
- Dose-finding Phase (Experimental): An initial group of 6 to 12 participants with cat allergy as defined by the eligibility criteria will undergo a single-visit, stepwise dose-escalating nasal allergen challenge only, with the aim of estimating the most appropriate single dose of allergen to use in the randomized phase. Eligible participants who participate in the dose-finding phase may proceed to the randomized phase of the trial after a minimum 28-day washout period.
  Interventions: Procedure: Nasal Allergen Challenge; Biological: Cat allergen (FelD1)

INTERVENTIONS:
Procedure: Nasal Allergen Challenge — Cat allergen (FelD1) applied directly to the nasal tissues
Other: Environmental Exposure Chamber — The mobile EEC (mEEC) is a movable facility, designed with clean-room technology, used to expose subjects to aeroallergens (in this trial, the allergen FelD1 from cats) at controlled, consistent airborne levels, similar to that experienced in subjects' daily lives.
  Other Names: EEC
  Arms: EEC Followed by NAC; NAC Followed by EEC
Biological: Cat allergen (FelD1)

SUMMARY:
This is a pilot trial in cat allergic participants, designed to compare allergic responses in each participant to a specific allergen by two methods of exposure. The methods of exposure to be used are: the environment exposure chamber (EEC) and nasal allergen challenge (NAC). Potential participants will be screened for evidence of cat allergy.

Participants with a range of allergic sensitivities to cat allergen will be enrolled. To help ensure some breadth in the level of allergic sensitivity among participants, individuals with both high and low exposures to cat allergens in their daily lives will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. History of moderate to severe allergic rhinitis (AR) caused by cat exposure for at least 2 years.
2. Skin prick test mean wheal diameter ≥ 5 mm larger than negative control to standardized cat extract at screening.
3. Non-pregnant, non-lactating women. For women of childbearing age, a willingness to use an effective form of contraception for the duration of the trial.
4. In general good health based on medical history and physical exam.
5. The ability to give informed consent and comply with study procedures.

Exclusion Criteria:

1. A history of anaphylaxis to cat allergen.
2. Prebronchodilator FEV1 less than 80% of predicted value at screening visit.
3. History of moderate/severe ARIA (Allergic Rhinitis and its Impact on Asthma) severity classification for allergic rhinitis for most of previous year in the absence of cat exposure (ARIA classification citation: Bousquet J, Khaltaev N, Cruz AA, et al. Allergy 2008; 63 Suppl 86:8-160.)
4. History of asthma symptoms or exacerbations in the past 12 months requiring regular inhaled corticosteroids for greater than 4 weeks per year, any oral corticosteroid usage, any emergency department visit for asthma or any asthma-related hospitalization.
5. Participants who, at the discretion of the investigator, suffer from seasonal allergic rhinitis to interfering allergens that cannot complete the study outside of the local pollen season or who have significant allergy to other perennial allergens that cannot be avoided during the study.
6. History of serious chronic medical conditions which might interfere with treatment or assessments or may pose additional risks from participation in the study.
7. History of chronic obstructive pulmonary disease (COPD).
8. History of significant recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment.
9. History of chronic sinusitis, defined as a sinus symptoms lasting greater than 12 weeks that includes 2 or more major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, and ear pain, pressure, or fullness.
10. History of systemic disease affecting the immune system such as autoimmune diseases, immune complex disease, or immunodeficiency, where, in the opinion of the study physician, participation in the trial would pose a risk or significant effect on the immune system.
11. Evidence of any active or suspected bacterial, viral, fungal or parasitic infections within 30 days prior to allergen challenge.
12. Exposure to an individual with active tuberculosis within six months prior to allergen challenge.
13. At time of allergen challenge, current symptoms of, or treatment for, an upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
14. History of cancer within the last 5 years, except for nonmelanoma skin cancer, stage 1 renal cell carcinoma, stage 1 prostate cancers cured by local resection and any curatively treated carcinomas in situ.
15. Any tobacco smoking within the last year or a history of ≥10 pack years.
16. Allergen immunotherapy treatment with cat within the previous 5 years.
17. Any history of grade 4 anaphylaxis due to any cause as defined by the CTCAE grading criteria.
18. History of bleeding disorders, treatment with anticoagulation or anti-platelet therapy or chronic treatment with aspirin for cardiovascular prophylaxis.
19. Treatment with omalizumab within 6 months prior to the NAC or EEC procedures.
20. Currently taking any of the following medications: beta blockers; tricyclic antidepressants; monoamine oxidase inhibitors.
21. Ongoing systemic immunosuppressive treatment.
22. History of intolerance to rescue medications or their excipients.
23. For women of childbearing age a positive urine pregnancy test with sensitivity of less than 50 mIU/mL.
24. The use of any investigational drug within 30 days of the NAC or EEC procedures.
25. The presence of any medical condition that the investigator deems incompatible with participation in the trial.
26. Any clinically significant abnormal finding on physical examination, vital signs or laboratory results at screening as deemed so by the Investigator.
27. Any clinically significant physical findings of nasal anatomical deformities (including the presence of nasal mucosal ulceration, nasal polyps, purulent secretions, septal perforation or any other major abnormalities in the nose) which, at the discretion of the Investigator, would interfere with the study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
NAC Total Nasal Symptom Score (TNSS) Area under the Curve (AUC) | Hour 0 to Hour 3 of Day 1 (for "NAC first" arm) or Day 30 (for "EEC first" arm)
  TNSS AUC evaluated from hour 0 to hour 3 of the NAC
EEC TNSS AUC | Hour 0 to Hour 3 of Day 2 (for "EEC first" arm) or Day 30 (for "NAC first" arm)
  TNSS AUC evaluated from hour 0 to hour 3 of the EEC

SECONDARY OUTCOMES:
TNSS AUC with NAC | Hour 0 to Hour 2
TNSS AUC with EEC | Hour 1 to Hour 3
  Recorded on second day of EEC.
Peak TNSS Score | Hour 0 to Hour 8
  Peak TNSS score during NAC and EEC.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Durham, MD, Study Chair — Imperial College London; Piyush Patel, MD, Principal Investigator — Inflamax Research Incorporated
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada

REFERENCES:
- [Background] Walker SM, Durham SR, Till SJ, Roberts G, Corrigan CJ, Leech SC, Krishna MT, Rajakulasingham RK, Williams A, Chantrell J, Dixon L, Frew AJ, Nasser SM; British Society for Allergy and Clinical Immunology. Immunotherapy for allergic rhinitis. Clin Exp Allergy. 2011 Sep;41(9):1177-200. doi: 10.1111/j.1365-2222.2011.03794.x. PMID 21848757
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org